CLINICAL TRIAL: NCT03761160
Title: Mobile Health App to Mitigate the Metabolic Effects of Androgen Deprivation Therapy: A Randomize Pilot Trial in Men Newly Treated With Androgen Deprivation Therapy
Brief Title: Mobile Health App to Mitigate the Metabolic Effects of Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Principal Investigator, Quoc-Dien Trinh, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-692
Record Dates: First submitted 2018-11-03; First posted 2018-12-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health App (Experimental): The developed mobile health app will include the following facets:
  * Physical activities
  * Dietary regimen.
  * The physical activities facet will encourage patients to engage in physical activities, with daily prompts, encouragement, and tips.
  * Users will be asked to record the type of physical activity they engaged in during the week, and for how long.
  * The dietary aspect will ask patients to log what they ate during the day and to rate how 'healthy' it is
  Interventions: Other: Mobile Health App
- Usual Care (Active Comparator): Usual care per hospital guideline
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Mobile Health App — mobile health app aims to provide patients who are about to initiate androgen deprivation therapy for prostate cancer with an exercise program and better eating habit
  Arms: Mobile Health App
Other: Usual care — Usual care per hospital guidelines
  Arms: Usual Care

SUMMARY:
This research study seeks to develop and evaluate a mobile health app which aims to provide patients who are about to initiate androgen deprivation therapy for prostate cancer with an exercise program and better eating habits.

DETAILED DESCRIPTION:
This research study seeks to develop and evaluate a mobile health app which aims to provide patients who are about to initiate androgen deprivation therapy for prostate cancer with an exercise program and better eating habits. The first phase of the research study seeks to evaluate the experience of the first version of the mobile health app within a group of participants and what they think of it.

The investigators are interested in how individuals react to the use of a developed mobile health app and what they think of it.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* All recruited participants must have owned a smartphone for >1 year
* English-speaking.
* Patients with prostate cancer aged between 40-75 years will be considered.
* No specific timeframe after prostate cancer diagnosis will be required for these patients.
* No limitations regarding their disease characteristics will be imposed (e.g. metastatic disease).
* Patients may or may not be currently receiving treatment Staff members will be recruited from
* Dana-Farber Cancer Institute Department of Medical Oncology,
* Brigham and Women's Hospital, Department of Surgery. Staff members aged between 40-75 years old will be considered. Phase 2
* Men diagnosed with prostate cancer presenting to DF/BWHCC
* About to initiate ADT for the first time will be considered.
* Age range 40-75-years
* The ability to walk 400 m
* Medical clearance from their primary physician
* English speaking
* Cognitively alert
* Literate
* Ability to read or hear with or without contacts/glass and hearing aid
* Ownership of a smartphone for >1yr

Exclusion Criteria:

* Men who have been under a rigorous structured exercise regime, such as individuals who engage in more than 900 minutes of moderate physical activity per week in the last 6 months will not be considered
* Post-ADT treatment
* Planned systemic chemotherapy
* Planned treatment with abiraterone or enzalutamide
* Bone metastases
* Acute illness
* Any musculoskeletal, cardiovascular, or neurologic disorders that could inhibit or put them at risk from exercising
* Subordinates to the PI

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Accumulation of body fat mass | 2 years
  This endpoint will be assessed with dual-energy x-ray absorptiometry - also known as a DEXA scan.

SECONDARY OUTCOMES:
Whole-body lean mass | 2 years
  This endpoint will be assessed with dual-energy x-ray absorptiometry - also known as a DEXA scan.
Regional lean mass | 2 years
  This endpoint will be assessed with dual-energy x-ray absorptiometry - also known as a DEXA scan.
Percent fat | 2 years
  This endpoint will be assessed with dual-energy x-ray absorptiometry - also known as a DEXA scan.
Estimated visceral adipose | 2 years
  This endpoint will be assessed with dual-energy x-ray absorptiometry - also known as a DEXA scan.
Application's performance on iOS and Android platforms | 2 years
  This outcome (for phase 1 of the trial) will be collected in 10 participants through verbal responses and/or computer either by the research coordinator or the participant. All data collected will be anonymously recorded.
Application's ability to effectively motivate and track outcomes for patients | 2 years
  This outcome (for phase 1 of the trial) will be collected in 10 participants through verbal responses and/or computer either by the research coordinator or the participant. All data collected will be anonymously recorded.

CONTACTS AND LOCATIONS:
Overall Officials: QUOC-DIEN TRINH, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].